CLINICAL TRIAL: NCT00350597
Title: Immunologic and Antibody Responses in Patients Receiving GM-CSF, (Leukine, Sargramostim) as Adjuvant Therapy of Stage II (T4), III and IV Melanoma.
Brief Title: GM-CSF as Adjuvant Therapy of Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northern California Melanoma Center (Other)
Collaborators: Bayer (Industry); Melanoma Research Institute (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GM-CSF 040906
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2006-07-11 (Estimated); Status verified 2006-07

CONDITIONS: Malignant Melanoma
Keywords: Malignant Melanoma; Adjuvant Therapy; Cytokine Therapy; Immunologic Testing
MeSH Terms: conditions — Melanoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

INTERVENTIONS:
Drug: Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF)

SUMMARY:
This is a pilot study to describe the immunological responses and clinical outcome associated with administration of recombinant human Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) as surgical adjuvant therapy in patients with malignant melanoma who are at high risk for recurrence (Stage II T4, III and IV).

DETAILED DESCRIPTION:
This is a pilot study to describe the immunological responses and clinical outcome associated with administration of recombinant human Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) as surgical adjuvant therapy in patients with malignant melanoma who are at high risk for recurrence (Stage II T4, III and IV). The immunological responses include serum neopterin levels. In a sub-set of study participants, additional immunologic testing will be done, including monocyte cytotoxicity to a melanoma cell line and phenotypic and functional markers of dendritic and T cell activation in peripheral blood mononuclear cells. The clinical end points of the study include safety, time to disease recurrence, time to disseminated disease, and survival. Eligible patients are those with high-risk melanoma who are clinically tumor free following surgery. Treatment will consist of GM-CSF at 125 g/m2 once daily (maximum dose 250 g) for 14 days followed by 14 days of rest (28 day cycle) for 1 year. Clinical status will be monitored until death or until the patient has been tumor free for five years, whichever event occurs first. Immunologic responses will be determined pretreatment, at the end of the first 14 days of dosing (Day 15), after the 14-day rest period (Day 29) and at the end of 14 days of dosing in cycles 6 (Day 155) and 13 (Day 351). Clinical outcome will be determined according to patient risk group (ultra-high risk Stage IIIC or IV versus high-risk Stage II T4, Stage IIIA and Stage IIIB). The pilot study will also assess the association of the immunological responses with clinical response and safety by patient risk group.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be males or females with histologically proven melanoma. Patients must have Stage II (T4), III, and IV malignant melanoma surgically resected with no clinical evidence of disease by clinical, laboratory criteria or radiologic examination as defined below.
* Individuals must be at least 14 years of age.
* Pregnant women are not eligible. Men and women will be required to use an effective form of contraception.
* Patients requiring corticosteroid therapy or are receiving other forms of immunotherapy are not eligible.
* Patients may have received immunotherapy for prior disease. They must have completed therapy at least one month prior to study entry. Patients may not have received prior chemotherapy or therapy with GM-CSF. Patients are permitted to receive adjuvant radiation therapy but these patients will not be selected as part of the sub-set undergoing studies of cellular immunologic responses since the radiation could alter these responses. Based on the reults from one randomized, controlled clinical trial, the LEUKINE product labeling contains the following contraindication: "Due to the potential sensitivity of rapidly dividing hematopoietic progenitor cells, LEUKINE should not be administered simultaneously with cytoxic chemotherapy or radiotherapy or within 24 hours preceding or following chemotherapy or radiotherapy. In one controlled study, patients with small cell lung cancer received LEUKINE and concurrent thoracic radiotherapy and chemotherapy or the identical radiotherapy and chemotherapy without LEUKINE. The patients randomized to LEUKINE had significantly higher incidence of adverse events, including higher mortality and a higher incidence of grade 4 infections and grade 3 or 4 thrombocytopenia.28" Other investigators have reported that CM-CSF can be given safely with concurrent radiation therapy. These contrasting results may be related to differences in the patient populations or intensity and/or location of the site of radiotherapy in the body, among other factors. GM-CSF has been administered safely in combination with radiation therapy for treatment of head and neck cancers29,30 and has been used safely during regimens that combine chemotherapy and radiation therapy.31
* Patients must undergo examination for evidence of residual disease, including physical examination, CBC, chemistry panel, CT scan of the chest and abdomen (and pelvis for lower extremity or lower trunk lesions), and single sequence with gadolinium MRI or CT of the brain. A PET scan may be substituted for the CT of the chest and abdomen (and pelvis). These tests must be negative for residual disease before entry into the study.
* Administration of the protocol medication must be initiated within 90 days of the definitive surgical excision rendering the patient NED.

Exclusion Criteria:

* Patients not meeting Inclusion Criteria described above

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2004-09; Study Completion 2010-07

PRIMARY OUTCOMES:
1 To describe the effect of GM-CSF adjuvant treatment of 125 ug/m2 once daily for 14 days followed by 14 days rest on immunological function as determined by serum neopterin levels (a measure of macrophage activation) and on serum levels of S100B.

SECONDARY OUTCOMES:
To evaluate if a change of any or all of the immunological parameters over the treatment period is associated with safety and/or clinical outcome as measured by time to disease recurrence, time to disseminated disease and/or survival.
To perform a more detailed immunologic analysis in a sub-set of study participants (6 evaluable patients) to determine the immunologic responses induced by GM-CSF. There are three main immunological analyses to be determined:
a Monocyte cell numbers and activity
b Mature dendritic cell numbers
c Surface markers on peripheral blood mononuclear cells (PBMC) relative to T cells

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E. Spitler, MD, Principal Investigator — Northern California Melanoma Center
Locations (1):
- Northern California Melanoma Center, San Francisco, California, United States

REFERENCES:
- [Background] Spitler LE, Grossbard ML, Ernstoff MS, Silver G, Jacobs M, Hayes FA, Soong SJ. Adjuvant therapy of stage III and IV malignant melanoma using granulocyte-macrophage colony-stimulating factor. J Clin Oncol. 2000 Apr;18(8):1614-21. doi: 10.1200/JCO.2000.18.8.1614. PMID 10764421
- See also: Northern California Melanoma Center Website — http://www.melanomacenter.com